CLINICAL TRIAL: NCT01258088
Title: A Randomized, Double-blind, Vehicle-controlled, Multiple Cohort Study To Determine The Safety, Tolerability, And Pharmacokinetic Profile Of An2728 Ointment B, 2% In Healthy Volunteers And Patients With Mild-to-moderate Plaque-type Psoriasis
Brief Title: Safety Study of Ointment for the Treatment of Plaque-type Psoriasis
Acronym: AN2728-PSR-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2728-PSR-104; C3291010 (Other: Alias Study Number)
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Plaque-type Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: AN2728 Ointment (Active Comparator)
  Interventions: Drug: AN2728 Ointment
- Cohort 1: AN2728 Vehicle (Placebo Comparator)
  Interventions: Drug: AN2728 Vehicle
- Cohort 3: AN2728 Ointment (Active Comparator)
  Interventions: Drug: AN2728 Ointment
- Cohort 3: AN2728 Vehicle (Placebo Comparator)
  Interventions: Drug: AN2728 Vehicle

INTERVENTIONS:
Drug: AN2728 Ointment — 5mg/cm2, BID
  Arms: Cohort 1: AN2728 Ointment; Cohort 3: AN2728 Ointment
Drug: AN2728 Vehicle — 5mg/cm2 BID
  Arms: Cohort 1: AN2728 Vehicle; Cohort 3: AN2728 Vehicle

SUMMARY:
The purpose of this study is to determine how much drug is absorbed throughout the body after being applied to the skin.

ELIGIBILITY:
Inclusion Criteria:

* White males, 18 - 55 years (inclusive) of age at the time of randomization.
* Body weight between 60-90 kg (Body Mass Index [BMI] between 19 and 30 kg/m2 [inclusive]).
* Willing and able to comply with study instructions and commit to all follow-up visits.
* Have adequate venous access to permit repeated PK sampling.
* Ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol-related procedures.
* Non-smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication).

For psoriasis patients (in addition to the above criteria):

* Clinical diagnosis of stable plaque-type psoriasis with active plaques involving 5%-20% of total BSA excluding face, scalp and groin.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug; or known allergy to any of the test product(s) or any components in the test product(s) or history of hypersensitivity; or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the Investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the distribution, metabolism or excretion of drugs.
* Abnormal physical findings of clinical significance at the Screening examination or Baseline which would interfere with the objectives of the study.
* History of orthostatic hypotension (an increase in HR ≥20 bpm accompanied by a ≥20 mm Hg drop in SBP and/or ≥10 mm Hg drop in DBP) present at Screening.
* Clinically significant abnormal laboratory values (as determined by the Investigator) at the Screening evaluation.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* 12-lead ECG obtained at Screening with: PR >240 msec, QRS >110 msec and QTc >450 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes on the Screening ECG, or any other changes on the Screening ECG that would interfere with measurement of the QT interval.
* Major surgical interventions within 6 months of the study.
* Has a positive pre-study Hepatitis B surface antigen; positive Hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV antibody result.
* Use of prescription or non-prescription drugs, including vitamin supplements, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 28 days prior to the first dose of study medication. However, the Investigator and study team can review medication use on a case by case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation. By exception, the subject may take paracetamol or acetaminophen (≤2 g/day) or ibuprofen (≤1600 mg/day) up to 48 h prior to the first dose of study medication.
* Has a history of regular alcohol consumption averaging >14 drinks/week (1 drink [100 mL wine or 280 mL standard strength beer or 30 mL of 80 proof distilled spirits]) within 6 months of the Screening visit.
* Loss of 500 mL blood or more during the 3 month period before the study, e.g., blood donor.
* People that follow vegetarian or vegan diets.
* Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
* History of drug abuse or dependence within 12 months of the study.
* Positive pre-study urine drug and alcohol screen. A minimum list of drugs that will be screened for include benzodiazepines, opiates, methadone metabolite (EDDP), sympathomimetic amines, cannabinoids, barbiturates, cocaine, and ethanol. (Suspected false positive results may be repeated at the discretion of the Investigator.)
* Concurrent or recent (within 60 days) participation in another drug or device research study.
* Considered by the Investigator to be unsuitable candidate for this study. Use of AN2728 in a previous clinical trial.

For psoriasis patients (in addition to the above exclusion criteria):

* Spontaneously improving or rapidly deteriorating psoriatic plaques or pustular/exfoliative, guttate, erythrodermic or other non-plaque form of psoriasis.
* Currently have drug-induced psoriasis (new onset or exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Other serious skin disorder(s).
* Use of non-biologic systemic anti-psoriatic therapy (e.g., corticosteroids, PUVA, UVB, retinoids, methotrexate, cyclosporine, other immunosuppressive agents) or biologic therapy (e.g., alefacept, etanercept, adalimumab, ustekinumab) within four weeks prior to enrollment or concurrently during the study.
* Use of topical treatments that have a known beneficial effect on psoriasis, including but not limited to corticosteroids, retinoids, vitamin D derivatives, tar or anthralin, within the past two weeks prior to enrollment or concurrently during the study.
* Systemic medications for other medical conditions that are known to affect psoriasis (e.g., lithium, beta adrenergic blockers) within the past four weeks prior to enrollment or concurrently during the study.
* Use of emollients/moisturizers on area(s) to be treated within two days prior to enrollment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2010-12-07 (Actual); Study Completion 2010-12-07 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 21 days
  12-lead ECG, clinical laboratory tests, urinalysis, spontaneous/elicited adverse event (AE) reporting, local site reactions, physical exam and vital signs (blood pressure, heart rate).

SECONDARY OUTCOMES:
Pharmacokinetic profile | 16 Days Maximum
  Non-compartmental analysis of classic PK parameters: AUC(0-t), Cmax, Tmax, terminal t-1/2 (computed if data from majority of subjects permit) of AN2728, on Days 1 and 7 (or last day of administration). Trough plasma concentrations at the end of the dosing interval (Ctrough) collected at pre-morning dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Sepehr Shakib, MB BS, PhD, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- CMAX (A Division of IDT Australia Ltd), Adelaide, Australia